CLINICAL TRIAL: NCT01024556
Title: Observational Study With Additional Diagnostic Procedures on Anti-Tat Immune Response in HIV-1-infected HAART-treated Adult Subjects
Brief Title: Observational Study on Anti-Tat Immune Response in HIV-1-infected HAART-treated Adult Subjects
Acronym: ISS OBS T-002
Status: Completed | Type: Observational
Sponsor: Barbara Ensoli, MD (Other)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PHD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Other Study IDs: ISS OBS T-002
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infection
Keywords: HIV, HAART
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, PBMCs
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study is designed as a prospective observational study directed at evaluating the frequency, magnitude, quality and persistence (primary endpoint) of the anti-Tat immune response in highly active antiretroviral therapy (HAART)-receiving HIV-1 infected individuals, and to prospectively evaluate the immunological, virological and clinical outcome of anti-Tat positive versus anti-Tat negative subjects under successful HAART (secondary endpoint), in order to determine the impact of anti-Tat immunity on HIV disease progression as well as the potential use of anti-Tat immune response assessment for the clinical and therapeutic management of HAART-treated infected patients. This survey provided important information for the design, planning and conduction of future therapeutic vaccine trials based on the HIV-1 Tat protein in HAART-treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV-1 infection
* To be under successful HAART treatment with plasma viremia <50 copies/ml in the last 6 months prior to initiation of the study, without a history of virologic rebound
* Known CD4+ T cells nadir
* Age ≥ 18 years old
* Signed informed consent

Exclusion Criteria:

* Current therapy with immunomodulators or immunosuppressive drugs, or chemotherapy for neoplastic disorders
* Concomitant treatment for HBV or HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hiv-1-infected haart-treated adult subjects
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2008-03; Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assessment of anti-Tat antibodies in sera of subjects, and of the proliferative response (CFSE) and the production of γIFN, IL-4 and IL-2 (Elispot) by peripheral blood mononuclear cells (PBMC) in response to Tat.

SECONDARY OUTCOMES:
The decline of CD4+ T cell counts, the increase of HIV plasma viral load or the occurrence of AIDS-defining events were assessed to determine progression to disease.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Esposito, MD, Principal Investigator — Azienda Ospedaliero - Universitaria Policlinico di Modena, Modena, Italy; Giovanni Di Perri, MD, Principal Investigator — Amedeo di Savoia Hospital, Turin, Italy; Adriano Lazzarin, MD, Principal Investigator — San Raffaele Hospital - Milan, Italy; Massimo Galli, MD, Principal Investigator — L. Sacco Hospital- Milan, Italy; Giampiero Carosi, MD, Principal Investigator — "Spedali Civili" di Brescia , Brescia, Italy; Florio Ghinelli, MD, Principal Investigator — Azienda Ospedaliero - Universitaria di Ferrara, Ferrara, Italy; Francesco Mazzotta, MD, Principal Investigator — S. M. Annunziata Hospital, Florence, Italy; Guido Palamara, MD, Principal Investigator — S. Gallicano Hospital- Rome, Italy; Fabrizio Soscia, MD, Principal Investigator — S. M. Goretti Hospital- Latina, Italy; Giuseppe Pastore, MD, Principal Investigator — "Ospedale Policlinico Consorziale"-Bari, Italy
Locations (10):
- Italy (10):
  - S.M. Goretti Hospital, Latina, Rome
  - General Hospital of Bari, Bari
  - Spedali Civili di Brescia, Brescia
  - General Hospital-University of Ferrara, Ferrara
  - A.M. Annunziata Hospital, Florence
  - L. Sacco Hospital, Milan
  - San Raffaele Hospital, Milan
  - General Hospital-University of Modena, Modena
  - San Gallicano Hospital, Rome
  - Amedeo di Savoia Hospital, Torino

REFERENCES:
- [Background] Andre P, Groettrup M, Klenerman P, de Giuli R, Booth BL Jr, Cerundolo V, Bonneville M, Jotereau F, Zinkernagel RM, Lotteau V. An inhibitor of HIV-1 protease modulates proteasome activity, antigen presentation, and T cell responses. Proc Natl Acad Sci U S A. 1998 Oct 27;95(22):13120-4. doi: 10.1073/pnas.95.22.13120. PMID 9789051
- [Background] Arya SK, Guo C, Josephs SF, Wong-Staal F. Trans-activator gene of human T-lymphotropic virus type III (HTLV-III). Science. 1985 Jul 5;229(4708):69-73. doi: 10.1126/science.2990040.
- [Background] Ensoli B, Barillari G, Salahuddin SZ, Gallo RC, Wong-Staal F. Tat protein of HIV-1 stimulates growth of cells derived from Kaposi's sarcoma lesions of AIDS patients. Nature. 1990 May 3;345(6270):84-6. doi: 10.1038/345084a0. PMID 2184372
- [Background] Ensoli B, Buonaguro L, Barillari G, Fiorelli V, Gendelman R, Morgan RA, Wingfield P, Gallo RC. Release, uptake, and effects of extracellular human immunodeficiency virus type 1 Tat protein on cell growth and viral transactivation. J Virol. 1993 Jan;67(1):277-87. doi: 10.1128/JVI.67.1.277-287.1993. PMID 8416373
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Monini P, Cafaro A, Srivastava IK, Moretti S, Sharma VA, Andreini C, Chiozzini C, Ferrantelli F, Cossut MR, Tripiciano A, Nappi F, Longo O, Bellino S, Picconi O, Fanales-Belasio E, Borsetti A, Toschi E, Schiavoni I, Bacigalupo I, Kan E, Sernicola L, Maggiorella MT, Montin K, Porcu M, Leone P, Leone P, Collacchi B, Palladino C, Ridolfi B, Falchi M, Macchia I, Ulmer JB, Butto S, Sgadari C, Magnani M, Federico MP, Titti F, Banci L, Dallocchio F, Rappuoli R, Ensoli F, Barnett SW, Garaci E, Ensoli B. HIV-1 tat promotes integrin-mediated HIV transmission to dendritic cells by binding Env spikes and competes neutralization by anti-HIV antibodies. PLoS One. 2012;7(11):e48781. doi: 10.1371/journal.pone.0048781. Epub 2012 Nov 13. PMID 23152803
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Background] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- [Result] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Derived] Tripiciano A, Picconi O, Moretti S, Sgadari C, Cafaro A, Francavilla V, Arancio A, Paniccia G, Campagna M, Pavone-Cossut MR, Sighinolfi L, Latini A, Mercurio VS, Pietro MD, Castelli F, Saracino A, Mussini C, Perri GD, Galli M, Nozza S, Ensoli F, Monini P, Ensoli B. Anti-Tat immunity defines CD4+ T-cell dynamics in people living with HIV on long-term cART. EBioMedicine. 2021 Apr;66:103306. doi: 10.1016/j.ebiom.2021.103306. Epub 2021 Apr 7. PMID 33839064
- See also: Related Info — http://www.hiv1tat-vaccines.info